CLINICAL TRIAL: NCT02656082
Title: A Single Arm, Phase II Open Label Trial to Investigate the Efficacy and Safety of Intra-dermal Injection of Etanercept for Remission Induction in Discoid Lupus Erythematosus
Brief Title: Targeted Therapy Using Intradermal Injection of Etanercept for Remission Induction in Discoid Lupus Erythematosus
Acronym: TARGET-DLE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Leeds (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); Pfizer (Industry); Clinical Trials Research Unit, Leeds (Unknown)
Responsible Party: Principal Investigator, Yuzaiful Md Yusof, Principal Investigator, University of Leeds
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RR15/114; 2015-001602-33 (EudraCT Number)
Record Dates: First submitted 2016-01-08; First posted 2016-01-14 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Lupus Erythematosus, Discoid; Lupus Erythematosus, Cutaneous; Lupus Erythematosus, Chronic Cutaneous
Keywords: Discoid lupus erythematosus; Intradermal injection of etanercept
MeSH Terms: conditions — Lupus Erythematosus, Discoid; Lupus Erythematosus, Cutaneous | interventions — Etanercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Etanercept (Experimental): Intradermal injection of etanercept. The dosage is determined based on discoid lesion radius. Weekly injection up to 12 weeks.
  Interventions: Drug: Etanercept

INTERVENTIONS:
Drug: Etanercept — Treatment with etanercept is intended for remission induction of DLE only and not for maintenance purpose.
  Other Names: Enbrel

SUMMARY:
The purpose of this study is to determine whether Etanercept which is given through intradermal injection is effective in the treatment of discoid lupus erythematosus (DLE).

The investigators also would like to develop new tests to measure skin inflammation by scanning the affected skin using optical coherence tomography (OCT), thermography and laser doppler imaging (LDI) and taking photographs of the rash (to be done before and after treatment). If the findings from these new tests are similar to the ones from taking a sample of skin (biopsy), then the latter (which is an invasive test) can be avoided.

DETAILED DESCRIPTION:
There is an unmet need for new therapies to control inflammation in discoid lupus erythematosus (DLE). A significant proportion of DLE patients (with or without systemic lupus erythematosus (SLE)) are resistant to conventional therapies and DLE may be exacerbated by B cell depletion therapy.There is no clinical guideline or algorithm on how to manage patients with DLE who have refractory disease to the first line agents, anti-malarials. If left untreated, uncontrolled inflammation will lead to permanent disfiguring and irreversible scar to the patient, thus pose a major cosmetic issue and significantly impair the quality of life.

Targeted therapy based on immunopathogenesis is an attractive approach and tumour necrosis factor (TNF) is implicated in the pathogenesis of DLE. However, systemic administration of TNF blockers has been associated with induction of pathogenic autoantibodies that may render SLE worse or progression from DLE only to SLE. TNF blockers have been administered using the intra-dermal injection route in other TNF-mediated diseases and appear similarly safe and effective to systemic administration.

Another issue is the problem with outcome measures as skin disease is particularly heterogenous and many instruments rely on subjective assessment which may be difficult even in the hands of experts.

The TARGET-DLE trial will address these problems by: (i) administering a TNF blocker, etanercept using the intra-dermal route, which will provide local concentration to neutralise TNF in tissue while minimises the effect to systemic immunity and (ii) measuring tissue response using the existing outcome measure; the modified limited Score of Activity and Damage in DLE (SADDLE) as well as new objective measures such as skin biopsy, optical coherence tomography (OCT), thermography and laser Doppler imaging (LDI).

Data from this study may be used to power a definitive randomised controlled trial should the primary end point be achieved.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-80 years old.
* Have at least one active DLE lesion, either diagnosed by skin biopsy or confirmation by Dermatologist/ Rheumatologist.
* Patients with DLE only and SLE patients with DLE are included.
* Have refractory disease to an anti-malarial for at least 3 months as assessed by Dermatologist/Rheumatologist.
* Patients receiving anti-malarials must have been receiving them for at least 3 months prior to Screening, with a stable dose regimen for at least 28 days (±1 day) prior to Baseline (the first study drug administration)
* Ability to provide an informed consent.
* All male and female patients biologically capable of having children must agree to use a reliable method of contraception for the duration of the study and for a period of 3 weeks after their final dose of study drug. Acceptable methods of contraception are surgical sterilisation, oral, implantable or injectable hormonal methods, intrauterine devices or barrier contraceptives.

Exclusion Criteria:

* Any prior treatment with TNF-blockade therapies.
* Intramuscular or intra-dermal corticosteroid within 28 days of the Screening visit.
* Corticosteroid of greater than 10mg prednisolone daily equivalent, or change in oral steroid dose within 28 days prior to Baseline Visit.
* A change in the dose of other immunosuppressant including methotrexate, azathioprine and mycophenolate mofetil within 28 days (±1 day) prior to Baseline Visit.
* Concomitant therapies with any alkylating agents (e.g. cyclophosphamide, chlorambucil), other immunosuppressant including sulfasalazine and leflunomide, other biological agent particularly anakinra and abatacept and other experimental drug. If patients are on any of these, they need to be off therapies for at least 28 days prior to Baseline Visit to allow for washout.
* Evidence of an immunosuppressive state, including an active HIV infection, agammaglobulinaemias, T-cell deficiencies or Human T cell Lymphotrophic Virus Type 1 (HTLV-1).
* Chronic active infection such as hepatitis B or hepatitis C and tuberculosis. Patients with latent tuberculosis may be included if treated with chemoprophylaxis for at least 2 months before starting the study and to continue chemoprophylaxis for a total of 6 months.
* History of cancer within the last 5 years except for squamous or basal cell skin carcinoma that has been completely excised and treated cervical carcinoma in situ.
* Demyelinating diseases.
* Moderate to severe heart failure based on New York Heart Association (NYHA) functional class III and IV.
* Pregnancy.
* Breastfeeding.
* Planned surgery within the study period which is expected to require omission of study medication of 28 days or more.
* Receipt of live attenuated vaccine within 28 days prior to the Baseline Visit.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
The proportion of patients who achieve a reduction in the modified limited Score of Activity and Damage in Discoid Lupus Erythematosus (SADDLE) score by 20% of the baseline score in the index lesion | At Week 12
  A modified SADDLE score will be used; limited to only one index lesion and the efficacy is judged based on total score in activity component only.

SECONDARY OUTCOMES:
Change in Physician's Visual Analogue Scale (VAS) for global assessment of disease activity from Baseline | At Week 12
  The investigator will rate the overall disease activity status of the participant with respect to the DLE signs and symptoms and the functional capacity of the participant, using a 100mm VAS where 0 is "very good, asymptomatic, and no limitation of normal activities" and 100 is "very poor, very severe symptoms which are intolerable, and inability to carry out all normal activities."
Change in daily oral prednisolone dose from Baseline | At Week 12
  Corticosteroid doses should be converted to prednisolone-equivalent doses (if not taking prednisolone form of corticosteroid) for data analysis. Expressed in milligram (mg).
Change in Dermatology Life Quality Index (DLQI) from Baseline | At Week 12
  This participant-reported outcome consists of 10 questions concerning participants' perception of the impact of skin diseases on different aspects of their health related quality of life over the preceding week.
Change in Participant's VAS for global health assessment from Baseline | At Week 12
  Participants will rate their global assessment of their DLE disease activity for the day of the visit using a 100mm VAS where 0 is "very good, no symptoms" and 100 is "very poor, very severe symptoms."
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | From Baseline to 15 weeks
Number of participants with new development or worsening of positive anti-nuclear antigen (ANA) titres from Baseline | At Week 7 and 15
Number of participants with new development or worsening of positive anti-double stranded deoxyribonucleic acid (dsDNA) titres from Baseline | At Week 7 and 15
Number of participants with new development or worsening of positive anti-extract nuclear antigen (ENA) titres from Baseline | At Week 7 and 15
Number of participants with new development or worsening of positive anti-cardiolipin antibody (ACA) titres from Baseline | At Week 7 and 15
Change in complement (C3 and C4) levels below the normal limit (if normal at baseline) | At Week 7 and 15
Number of participants with detectable serum etanercept level | At Week 5
Change in disease activity as assessed using the British Isles Lupus Activity Groups (BILAG)-2004 score from Baseline | At Week 7 and 15
  This is only assessed in participants with systemic lupus erythematosus (SLE) rather than DLE only at Baseline
Change in disease activity as assessed using SLE Disease Activity Index (SLEDAI) from Baseline | At Week 7 and 15
  This is only assessed in participants with systemic lupus erythematosus (SLE) rather than DLE only at Baseline
Change in total histiopathologic score of skin biopsy from Baseline | At Week 12
  The skin biopsy will be scored for the classic histological features of DLE including (i) interface dermatitis (ii) vacuolar alteration of the basal layer, (iii) thickening of the basement membrane, (iv) follicular plugging, (v) hyperkeratosis, (vi) atrophy of the epidermis, (vii) inflammatory cell infiltrate in a perivascular, periappendageal and subepidermal location and (viii) dermal mucin deposition using a graded scale of 0-3; 0=none, 1=slight, 2=moderate and 3=strong for each feature.
Change in total OCT score from Baseline | At Week 12
  The OCT will be scored for (i) thickening and disruption of the entrance signal (ii) thinning of layer below the entrance signal (iii) patchy hyporeflective zones in the epidermis and (iv) wide signal free cavities in the upper dermis using a graded scale of 0-3; 0=none, 1=slight, 2=moderate and 3=strong for each parameter
Change in the difference in temperature between active DLE and nonactive area as assessed using thermography from Baseline | At Week 12
  Thermography is a non-invasive technique that detects infrared radiation to provide an image of the temperature distribution across skin surface. The temperature will be measured in Celcius
Change in perfusion per unit blood flow as assessed using LDI from Baseline | At Week 12
  LDI is a non-invasive imaging modality that is used to monitor blood perfusion in dermal tissue. Based on the well-established Doppler principle, this beam collects back-scattered light without touching the tissue and generates colour-coded images of the spatial distribution of tissue perfusion. This is expressed in terms of arbitrary perfusion units (PU).
Change in photograph score from Baseline | At Week 12
  The index lesion will be photographed using macro digital camera. These images will then be scored by two dermatologists who will be blinded to the clinical status, for response to therapy using a graded scale of 1-5; 1=remission, 2=slight improvement, 3=no change in response, 4=slight worsening and 5=severe worsening.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Emery, MD FMedSci, Study Chair — University of Leeds
Locations (1):
- Leeds Institute of Rheumatic and Musculoskeletal Medicine, Chapel Allerton Hospital, Leeds, United Kingdom